CLINICAL TRIAL: NCT02372955
Title: Mechanistic Study of the Systolic Blood Pressure Lowering Effect of Dapagliflozin in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gulf Regional Research & Educational Services, LLC (Other)
Responsible Party: Principal Investigator, Thomas Giles, Medical Director, Gulf Regional Research & Educational Services, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESR-14-10022/D1690L00020
Record Dates: First submitted 2015-01-07; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dapagliflozin 10 mg daily (Experimental): dapagliflozin, 10 mg daily for 16 weeks
  Interventions: Drug: dapagliflozin
- glimpiride (Active Comparator): glimpiride 4 mg daily for 16 weeks
  Interventions: Drug: glimpiride

INTERVENTIONS:
Drug: dapagliflozin — subjects will be randomly assigned to receive dapagliflozin 10 mg daily
  Other Names: Farxiga
  Arms: dapagliflozin 10 mg daily
Drug: glimpiride — subjects will be randomly assigned to receive glimpiride 4 mg daily
  Other Names: Amaryl
  Arms: glimpiride

SUMMARY:
Dapagliflozin has been shown to lower clinic systolic and diastolic blood pressure in patients with type 2 diabetes mellitus. The exact mechanism(s) by which dapagliflozin lowers clinic SBP is unknown. The primary objective of the study is to determine the effect of dapagliflozin , 10 mg daily, on parameters of arterial stiffness: aPWV, augmentation index (AI), 24-hour blood pressure patterns, SBP, and pulse pressure. Urinary sodium excretion, and Intravascular volume status will be recorded. The study will involve 21 subjects for a duration of 16 weeks.

DETAILED DESCRIPTION:
Dapagliflozin has been shown to lower clinic systolic and diastolic blood pressure in patients with type 2 diabetes mellitus. In particular, the reduction in SBP is impressive. The effect on circadian patterns of blood pressure measured by ambulatory blood pressure monitoring has not been established. The exact mechanism(s) by which dapagliflozin lowers clinic SBP is not clear although there has been speculation that it is due to a decrease in intravascular volume secondary to the osmotic diuresis produced by the drug. However, SBP is dependent on both pulse volume and vascular stiffness (impedance to ejection).

Dapagliflozin may have a favorable effect on vascular stiffness by a reduction in blood glucose resulting in decreased proximal arterial collagen cross-linking due to non-enzymatic glycosylation of proteins.

Dapagliflozin may also have a favorable effect on vascular stiffness by increasing urinary sodium excretion. Dapagliflozin is a sodium/glucose co-transporter inhibitor and the effects on sodium excretion are not clear. Increased sodium intake is associated with an increase in vascular stiffness.

An increase in vascular stiffness has been correlated with increased cardiovascular morbidity and mortality. Thus, it is important to know if dapagliflozin has an effect on vascular stiffness.

The current "gold standard" for vascular stiffness is aortic pulse wave velocity (aPWV). Other measures of vascular stiffness include: systolic blood pressure, pulse pressure and augmentation index. Also, measurement of calculated central blood pressure provides information that may not be apparent from measurement of brachial blood pressure.

Measures of intravascular volume status include: body weight, jugular venous pressure, orthostatic changes in blood pressure and heart rate.

It is important to recognize that some oral anti-diabetic drugs, e.g. sulfonylurea's are associated with an increase in systemic arterial blood pressure.

Hypothesis

That treatment of type 2 diabetes mellitus with dapagliflozin will result in a decrease in arterial stiffness

Primary Objectives

The primary objective of the study is to determine the effect of dapagliflozin (Appendix A), 10 mg daily, on parameters of arterial stiffness: aPWV, augmentation index (AI), 24-hour blood pressure patterns, SBP, and pulse pressure.

Key Questions

* What effect will dapagliflozin have on measures of arterial stiffness?
* What effect will dapagliflozin have on central blood pressure?
* Will dapagliflozin lower BP over the 24-hour period and will the pattern of BP change?
* Will dapagliflozin increase sodium excretion for 16 weeks?
* What will be the effect of dapagliflozin on intravascular volume status at 16 weeks?

Secondary Objectives

* Urinary sodium excretion
* Intravascular volume status: jugular venous pressure, body weight, orthostatic change in BP and pulse rate

Treatment

All patients will receive a background treatment with metformin. After randomization (2:1) patients will receive dapagliflozin, 10 mg daily or glimpiride (Appendix B), 4 mg daily. The treatment period will last ;16 weeks.

For high risk subjects, dapagliflozin therapy will begin with 5 mg with up-titration at 2 weeks. High risk subjects are those prone to volume depletion and are identified by signs of hypovolemia, e.g. low venous pressure, and a low arteriasl blood pressure.

Subjects will also be closely monitored for the development of hypoglycemia. This risk will be minimized by not enrolling subjects taking insulin. Subjects will be made aware of the signs of hypotlycemia, e.g. sweating and palpitation, and will be instructed to treat with ingestion of sugar, particularly fructose in orange juice.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Metformin treatment

Exclusion Criteria:

* • Type 1 diabetes mellitus

  * Hgb A1c > 9
  * Advanced diabetic complications, e.g. diabetic renal disease (eGFR < 60 cc/min), heavy proteinuria, diabetic retinopathy, autonomic neuropathy
  * Pregnancy or unwilling to practice contraception.
  * Uncontrolled hypertension (SBP > 150 mm Hg; DBP > 100 mm Hg)
  * Chronic substance abusers
  * Carcinoma of the urinary bladder
  * Subjects deemed at risk for dehydration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure by ambulatory blood pressure monitoring (ABPM) | 16 weeks
arterial stiffness | 16 weeks
  arterial stiffness will be assessed by measuring aortic pulse wave velocity (aPWV) and augmentation index

SECONDARY OUTCOMES:
urinary sodium excretion | 16 weeks
composite intravascular volume status | 16 weeks
  jugular venous pressure, body weight, orthostatic change in BP and pulse rate

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Regional Research & Educational Services, LLC, Metairie, Louisiana, United States